CLINICAL TRIAL: NCT03898687
Title: Sentinel Node Localisation and Staging With Superparamagnetic Iron Oxide-enhanced MRI and Magtrace®/Sentimag® in Patients With Malignant Melanoma of the Extremities. The MAGMEN Feasibility Study
Brief Title: The Use of Magtrace®/Sentimag® in Sentinel Node Biopsy for Malignant Melanoma. The Magmen Study.
Acronym: MAGMEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Dimitrios Katsarelias, Principal investigator, Sahlgrenska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DNR 947-18
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Melanoma; Sentinel Lymph Node
Keywords: melanoma; Sentinel node; SPIO-MRI
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAGMEN arm (Other): Patients with melanoma of the extremities included in the protocol. SLNB will be performed with the addition of magtrace (SPIO) injection, 0.2 ml around previous scar. The patients will undergo MRI of the involved basin (Axilla-groin)and receive the SpIO injection the day before SLN biopsy. A separate SPIO MRI will be performed before the operation. All patients will receive all 3 methods for SLN identification as described in the protocol.
  Interventions: Device: SLN Biopsy with Magtrace®/Sentimag®

INTERVENTIONS:
Device: SLN Biopsy with Magtrace®/Sentimag® — Identification of SLN by means of Magtrace®/Sentimag® and SPIO-MRI

SUMMARY:
To evaluate the use of superparamagnetic iron oxide (Magtrace®) as a tracer in sentinel node biopsy in malignant melanoma of the extremities, and to evaluate the possible role of Magtrace®-MRI for staging.

Primary objective:

• To evaluate if Magtrace®/Sentimag® can be used to identify SN in malignant melanoma with the same diagnostically reliability as the currently used method of Technetium 99m and Patent blue.

Secondary objectives:

• To evaluate if Magtrace®-MRI can predict sentinel node status in melanoma. This is a feasibility phase I, interventional single arm study. All patients included in the study will receive the same management.

20 patients will be included in the study. An enrollment time of 6-12 months is expected.

Primary endpoint • To determine the detection rate of Magtrace®/Sentimag® in comparison to SNB using technetium and blue dye in patients with malignant melanoma of the extremities.

Secondary endpoint

• To evaluate Magtrace®-MRI sensitivity and specificity as a preoperative tool for staging in malignant melanoma.

DETAILED DESCRIPTION:
Background Sentinel node biopsy (SNB) is a well-established technique for nodal staging of malignant disease, including breast cancer and malignant melanoma. The sentinel node (SN) is the first lymph node to receive cancer cells in a given lymph node basin. The status of the SN is often the most important prognostic factor, and determines potential adjuvant therapy and follow-up. The SN is detected by injection of a radioactive isotope (Technetium 99m) and a blue dye around the tumour or the scar following primary resection. This is achieved by a lymphoscintigraphy which is usually performed the day before surgery which necessitates a nuclear medicine department. At the time of surgery, a blue dye (Patent blue) is injected at the same area prior to incision. Thereafter the SN is identified by a handheld gamma-probe and the dye which colours the sentinel node blue. The so called hot and blue lymph node is removed surgically and sent to pathology for staging.

The mortality of cutaneous malignant melanoma is high, especially when diagnosed in an advanced stage [4]. Accurate staging and prediction of outcome largely depend on the identification and examination of the SN. SNB is recommended in Sweden for melanomas with a Breslow thickness more than 1 mm. About 20% of SNs in patients with melanoma are positive, which affects follow-up and also potentially adjuvant therapies that recently have been approved.

SNB is a surgical technique with associated risk for complications, mainly seroma, infections and lymph-edema. If nodal status could be determined by imaging, the dissection of the sentinel node biopsy could be avoided. However, current imaging techniques, such as MRI, CT and ultrasound are not accurate enough to stage the lymph nodes preoperatively. Motomura et al. recently reported a technique where superparamagnetic iron-oxide (SPIO) is injected into the tumour in patients with breast cancer, followed by MRI scan. They found a 100% sensitivity and 96% specificity for node staging when being compared to SNB.

There has been an increasing interest in using SPIO for identifying the sentinel node in breast cancer and recent publications showed great accuracy when SPIO was used as the only tracer. The agent was injected intra tumoral or subcutaneously under the areola before surgery and the SN(s) was/were detected by use of a handheld probe (Sentimag, Endomagnetics Ltd). The Sentimag is a magnetometer, which measures the strength of the magnetic field created by the iron oxide particles in the SPIO. It is a handheld device that signals when it is close enough to a magnetic field. The method was compared for feasibility and sensitivity to the current method used for identifying the SN (Technetium and Patent blue) and it was found to be at least as reliable and accurate.

Concerning melanoma, the SPIO method has not been used except recently when the MELAMAG trial was published. SPIO was compared to blue dye and radioisotope for identification of sentinel node in clinically node negative patients with melanoma. 97.7% of patients had a sentinel node identified with the standard technique, whereas 95.3% were identified with the magnetic tracer.

In view of these results, using SPIO as the only tracer to identify the sentinel node, in melanoma patients, instead of the double technique, could also be feasible. This could also be combined to SPIO MRI before surgery so as to evaluate this as a non-interventional method. The primary aim of this study is to evaluate the detection rate of SPIO (Magtrace®) in patients with melanoma of the extremities compared to technetium and blue dye. The secondary aim is to evaluate the specificity and sensitivity of SPIO (Magtrace®)-MRI.

STUDY OBJECTIVES AND DESIGN Study Objectives Primary objective

• To evaluate if Magtrace®/Sentimag® can be used to identify SN in malignant melanoma with the same diagnostically reliability as the currently used method of Technetium 99m and Patent blue.

Secondary objectives To evaluate if Magtrace®-MRI can predict sentinel node status in melanoma.

Study design Patients diagnosed with malignant melanoma of the extremities being candidates for wide local excision and SNB, will be considered for enrollment. Patients should have a primary melanoma located to one extremity, without clinically suspected lymph nodes metastasis on palpation and be planned for a SNB. A total of 20 patients that complete the study will be included. The study will be presented both by verbal and written means by one of the investigators. If the patient accepts enrolment, a written informed consent will be signed by both parties.

Patients will undergo an MRI of the lymph node basin (axillary or inguinal). Then they will receive an interstitial injection of Magtrace® with or without local anaesthesia up to a total of 2 ml divided in 4 doses injected in 4 quadrants around the previous excision scar. Care shall be taken for the injection not to exceed the excision area and thus cause a permanent skin discoloration after the wide local excision. After a minimum of 2 hours a new MRI (Magtrace®-MRI) of the same lymph node basin will be performed. The surgery will be scheduled within 7 days from the Magtrace® injection. The results of the Magtrace®-MRI will be evaluated to decide potential SNs and their status with the radiologist prior to surgery. The SN will be considered non-metastatic (negative) if it shows homogenous, low intensity signal on T2 weighted images compared to pre- Magtrace® images. A node will be considered as metastatic (positive) if the whole node or parts of it does not show a low intensity signal on T2 weighted image or if there is a high signal on water excitation compared to pre- Magtrace® images.All SNs identified by MRI will be considered for excision if they can be identified by using the Sentimag® probe.

A lymphoscintigraphy with Technetium-99m will be performed the day before surgery, in accordance to our current practice. Results will be investigated thoroughly and compared to the Magtrace®-MRI results, in order to identify discrepancies between the two methods.

During surgery, the current double technique, with the gamma probe and the blue dye, will be combined with the Sentimag, Endomagnetics Ltd probe and the intraoperative findings will be registered and analysed by the investigators, so as to test the feasibility of the method in comparison to the double method. All the nodes harvested will be sent to pathology and the final results will be compared to the Magtrace®-MRI results prior to surgery. CRF will be completed at the end of surgery and then when definitive pathology report is available. Data from all 20 patients included in this trial will be analysed at the end of the study. Patients will be followed according to clinical routine, no specific follow-up is required for this study.

ELIGIBILITY:
Inclusion Criteria:

A patient meeting ALL of the following criteria is eligible for participation in the study

1. Male or female aged above 18 years.
2. Signed and dated written informed consent before the start of specific protocol procedures.
3. Histologically confirmed melanoma of the extremities that is candidate to wide local excision and sentinel node biopsy (SLNB).
4. ECOG performance status 0-2

Exclusion Criteria:

A patient meeting ANY of the following criteria is not eligible for study participation:

1. Life expectancy of less than 6 months
2. Pregnant or breast-feeding.
3. Body Mass Index (BMI) > 45
4. Pacemaker or metal implants
5. Claustrophobia
6. Clinically suspect lymph nodes metastasis on palpation
7. Iron overload disease
8. Known hypersensitivity to iron or dextran compounds
9. Inability to understand given information and give informed consent or undergo study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Identification of Sentinel node with Magtrace®/Sentimag® | 12 months
  More than 95% success rate for identification of the Sentinel node with Magtrace®/Sentimag®

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Katsarelias, MD,Phd, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No